CLINICAL TRIAL: NCT07082725
Title: 18-month Double-blind, Randomized, Placebo-controlled, Multicenter, Phase 3 Study to Evaluate the Safety and Efficacy of Oral Nizubaglustat (AZ-3102) in Late-infantile and Juvenile Forms of Niemann-Pick Type C Disease and in Late-infantile and Juvenile-onset Forms of GM1 Gangliosidosis or GM2 Gangliosidosis
Brief Title: A Study to Evaluate the Safety and Efficacy of Oral Nizubaglustat (AZ-3102) in Late-infantile and Juvenile Forms of Niemann-Pick Type C Disease (NPC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Azafaros A.G. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZA-001-301-NPC; 2024-515778-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-27; First posted 2025-07-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Niemann-Pick Type C Disease
Keywords: Nizubaglustat
MeSH Terms: conditions — Niemann-Pick Disease, Type C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nizubaglustat (Experimental): Once daily oral dispersible tablets
  Interventions: Drug: Nizubaglustat
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nizubaglustat — AZ-3102
  Arms: Nizubaglustat
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
An 18-month double-blind, randomized, placebo-controlled, multicenter, Phase 3 study to evaluate the safety and efficacy of oral nizubaglustat (AZ-3102) in late-infantile and juvenile forms of Niemann-Pick type C disease

DETAILED DESCRIPTION:
Please see NCT #07054515 for information on the AZA-001-301 Master Protocol

PRIMARY OBJECTIVE

The primary objective of this study is to demonstrate superior efficacy on ataxic manifestations with oral nizubaglustat dosing compared with placebo when administered over 18 months in participants with late-infantile and juvenile forms of NPC disease

SECONDARY OBJECTIVES

I. To assess additional efficacy in ataxic and non-ataxic manifestations comparing nizubaglustat dosing with placebo when administered over 18 months in participants with late-infantile and juvenile forms of NPC disease

II. To assess the pharmacokinetic (PK) properties of nizubaglustat after administration of the first dose (Visit 1) and at steady state after multiple once daily doses

III. To assess the pharmacodynamic (PD) effects of nizubaglustat

IV. To assess the safety and tolerability of daily oral nizubaglustat dosing compared with placebo, when administered over 18 months in participants with late-infantile and juvenile forms of NPC disease

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Confirmed diagnosis of NPC disease
* Patient is unable or unwilling to take miglustat, or is, in the opinion of the investigator, unsatisfactorily treated with miglustat
* Male and female participants aged 4 years and older at the time of informed consent
* Onset of neurological symptoms from 2 to 15 years
* Disability level at Baseline: Ataxic disturbances with a total SARA score of ≥3 and ≤30 at Baseline
* Female of childbearing potential who are sexually active willing to follow the contraceptive guidance
* Male participants with a female partner of childbearing potential willing to follow the contraceptive guidance

Exclusion Criteria:

* A history of medical conditions other than NPC disease that, in the opinion of the Principal Investigator, would confound scientific rigor or the interpretation of results
* Body weight of <10 kg
* The presence of another neurologic disease
* The presence of moderate or severe hepatic impairment
* The presence of moderate or severe renal impairment
* Platelet count of <100x10^9/L
* The dose of any anti-epileptic treatment(s) was not stable (required a change in dose within the previous 3 months) and/or a new anti-epileptic treatment (drug or procedure) was prescribed in the month before Baseline
* Prior use of an investigational drug within the 3 months before Screening; or prior participation in a clinical study involving gene therapy or stem cell transplantation within 2 years prior to Screening
* A positive serum pregnancy test (for women of childbearing potential)
* Current treatment with miglustat, provided the patient has been using the recommended dose for most of the past 12 months AND is, in the opinion of the investigator, satisfactorily treated with miglustat. Any participants receiving miglustat are required to undergo a 1-month washout period before starting study medication

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-11-04 (Estimated); Study Completion 2027-11-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in total Scale for the Assessment and Rating of Ataxia (SARA) score | Baseline to month 18
  Total SARA comprises eight categories with a cumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia)
Change from baseline in functional SARA score | Baseline to month 18
  Functional SARA uses an abbreviated scale that scores 0 to 16, with higher scores indicating more severe impairment

SECONDARY OUTCOMES:
Change from baseline in SARA score for gait/posture | Baseline to months 6, 12, and 18
  Assessed on a 9-point scale with higher scores indicating inability to complete the task
Change from baseline in SARA score for speech | Baseline to months 6, 12, and 18
  Assessed on a 7-point scale with higher scores indicating unintelligible speech/anarthria
Change from baseline in SARA score for kinetics | Baseline to months 6, 12, and 18
  Assessed on a 5-point scale with higher scores indicating more severe impairment
Change from baseline in Vineland Adaptive Behavior Scale (VABS) | Baseline to months 6, 12, and 18
  Assesses four domains of function: communication, daily living skills, socialization, and motor skills
Change from baseline in Penetration-Aspiration Scale (PAS) | Baseline to months 6, 12, and 18
  Assessed on an 8-point ordinal scale, with 1 representing the lowest and 8 the highest/most severe score
Change from baseline in 9-Hole Peg Test (9-HPT-D) | Baseline to months 6, 12, and 18
  Assessed by the number of pegs per second placed in a 50-second, 9-HPT using the dominant hand
Change from baseline in NPC-Clinical Severity Scale (NPC-CSS) | Baseline to months 6, 12, and 18
  Scores can range from 0 to 61, with a higher score indicating more severe clinical impairment
Change from baseline in Goal Attainment scale (GAS) | Baseline to months 6, 12, and 18
  Assesses individual goals achieved during the study
Change from baseline in Clinician Global Impression of Change (CGI-C) | Baseline to months 6, 12, and 18
  Assessed on a 7-point scale with higher scores indicating lower improvement
Change from baseline in Participant/Caregiver Global Impression of Change (PGI-C) | Baseline to months 6, 12, and 18
  Assessed on a 7-point scale with higher scores indicating lower improvement
Change from baseline in Seizure frequency and duration, as per the seizure diary | Baseline to months 6, 12, and 18
Time-to-event comparison between nizubaglustat and placebo over the study duration for pre-defined detrimental events of an increase in total SARA score of ≥2 points | Baseline to month 18
Time-to-event comparison between nizubaglustat and placebo over the study duration for pre-defined detrimental events of an increase in functional SARA of ≥1.5 points | Baseline to month 18
Time-to-event comparison between nizubaglustat and placebo over the study duration for pre-defined detrimental events of a decrease in PAS of ≥1 point | Baseline to month 18
Time-to-event comparison between nizubaglustat and placebo over the study duration for pre-defined detrimental events of participants leaving the study due to participant/caregiver perception of disease progression/lack of efficacy | Baseline to month 18
Maximum observed plasma concentration (Cmax) | Baseline and months 1,18, and 21
Time to Cmax (Tmax) | Baseline and months 1,18, and 21
Plasma trough concentration (Ctrough) | Baseline and month 1
Area under the plasma concentration-time curve from time of dosing (zero) to 24 hours post-dose (AUC0-24) at baseline | Baseline (Day 1)
Accumulation ratio for Cmax | Baseline and months 1,18, and 21
Change from baseline in plasma concentration of glucosylceramide (GlcCer) C16:0; C18:0 | Baseline and months 1, 6, 12, and 18

CONTACTS AND LOCATIONS:
Locations (30):
- United States (4):
  - UCSF Children's Hospital and Research Center at Oakland, Oakland, California
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Children's Medical Center Dallas, Dallas, Texas
  - Lysosomal Rare Disorders Research and Treatment Center, Fairfax, Virginia
- Argentina (2):
  - Hospital Universitario Austral, Ciudad Autónoma Buenos Aires, Buenos Aires
  - Hospital de Niños de La Santisima Trinidad, Córdoba, Córdoba Province
- Australia (3):
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Children's Hospital Melbourne - PIN, Parkville, Victoria
- Brazil (3):
  - Instituto Fernandes Figueira, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul
  - Hospital Pequeno Principe, Curitiba
- Canada (3):
  - M.A.G.I.C. Clinic Ltd. Metabolics and Genetics in Calgary, Calgary, Alberta
  - University of Alberta Medical Genetics Clinic, Edmonton, Alberta
  - Centre Hospitalier de l'Universite de Montreal-1000 rue Saint-Denis, Montreal, Quebec
- SphinCS GmbH, Höchheim, Germany
- India (3):
  - Amrita Institute of Medical Sciences and Research Centre, Ernākulam, Kerala
  - All India Institute of Medical Sciences (AIIMS) - New Delhi, New Delhi, National Capital Territory of Delhi
  - JK Lone Hospital, Jaipur, Rajasthan
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy
- ULS de Santo António, EPE - Centro Materno Infantil Norte, Porto, Porto District, Portugal
- Spain (2):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona, Barcelona
  - Hospital Infantil Universitario Niño Jesus - PIN, Madrid, Madrid
- Inselspital - Universitätsspital Bern, Bern, Canton of Bern, Switzerland
- Turkey (Türkiye) (3):
  - Balcali Hastanesi Saglik Uygulama ve Arastirma Merkezi, Adana, Adana
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi, Çankaya, Ankara
  - Ege Universitesi Tip Fakultesi, Bornova, İzmir
- United Kingdom (3):
  - Great Ormond Street Hospital, London, London
  - University College London Hospitals (UCLH), London, Middlesex
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No